CLINICAL TRIAL: NCT01478321
Title: A Phase II Study of the Efficacy of Hypofractionated Radiation Therapy With Bevacizumab and Temozolomide Followed by Maintenance Temozolomide and Bevacizumab for Recurrent High-Grade Gliomas
Brief Title: Efficacy of Hypofractionated XRT w/Bev. + Temozolomide for Recurrent Gliomas
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual to some cohorts
Sponsor: Northwestern University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NU 11C02; STU00053636 (Other: Northwestern University IRB); NCI CTRP# (Other: NCI-2011-02904)
Record Dates: First submitted 2011-11-17; First posted 2011-11-23 (Estimated); Results first posted 2020-03-12 (Actual); Last update posted 2020-03-12 (Actual); Status verified 2019-07

CONDITIONS: Adult Anaplastic Astrocytoma; Adult Anaplastic Ependymoma; Adult Anaplastic Oligodendroglioma; Adult Giant Cell Glioblastoma; Adult Glioblastoma
Keywords: Information Not Provided
MeSH Terms: conditions — Astrocytoma; Ependymoma; Oligodendroglioma; Glioblastoma | interventions — Temozolomide; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (radiation, chemotherapy, monoclonal antibody) (Experimental): CONCURRENT THERAPY: Patients undergo hypofractionated radiation therapy 5 days a week beginning on day 0. Patients also receive temozolomide PO QD and bevacizumab IV over 30-90 minutes once every 2 weeks beginning on days -3 to 0. Treatment continues for 5 weeks in the absence of disease progression or unacceptable toxicity.
  ADJUVANT THERAPY: Beginning 2 weeks after completion of radiation therapy, patients receive temozolomide PO QD for 6 weeks and bevacizumab IV over 30-90 minutes once every 2 weeks. Courses repeat every 8 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Temozolomide; Radiation: hypofractionated radiation therapy; Biological: bevacizumab; Other: questionnaire administration

INTERVENTIONS:
Drug: Temozolomide — Given PO
  Other Names: TMZ
Radiation: hypofractionated radiation therapy — Undergo hypofractionated radiation therapy
Biological: bevacizumab — Given IV
  Other Names: anti-VEGF humanized monoclonal antibody,
Other: questionnaire administration — Ancillary studies

SUMMARY:
This phase II trial studies how well giving hypofractionated radiation therapy together with temozolomide and bevacizumab works in treating patients with high-grade glioblastoma multiforme or anaplastic glioma. Specialized radiation therapy, such as hypofractionated radiation therapy, that delivers a high dose of radiation directly to the tumor may kill more tumor cells and cause less damage to normal tissue. Drugs used in chemotherapy, such as temozolomide, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some block the ability of tumor to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Giving hypofractionated radiation therapy together with temozolomide and bevacizumab may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the overall survival (OS) for patients with recurrent high grade malignant gliomas treated with concurrent radiation, temozolomide, and bevacizumab followed by adjuvant temozolomide and bevacizumab.

SECONDARY OBJECTIVES:

I. Determine the impact of this regimen on neurologic symptoms via Functional Assessment of Cancer Therapy-Brain (FACT-Br) and FACT-Fatigue scales and Eastern Cooperative Oncology Group (ECOG) performance status.

II. Determine the safety profile of this regimen. III. Determine the progression free survival (PFS) at 6 and 12 months (all patients) as well as at 3 months (bevacizumab-exposed patients only).

OUTLINE:

CONCURRENT THERAPY: Patients undergo hypofractionated radiation therapy 5 days a week beginning on day 0. Patients also receive temozolomide orally (PO) once daily (QD) and bevacizumab intravenously (IV) over 30-90 minutes once every 2 weeks beginning on days -3 to 0. Treatment continues for 5 weeks in the absence of disease progression or unacceptable toxicity.

ADJUVANT THERAPY: Beginning 2 weeks after completion of radiation therapy, patients receive temozolomide PO QD for 6 weeks and bevacizumab IV over 30-90 minutes once every 2 weeks. Courses repeat every 8 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 2-3 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed diagnosis of glioblastoma multiforme (GBM) or anaplastic glioma, World Health Organization (WHO) grade 3 or 4

  * Patients must have measurable or non-measurable (evaluable) disease recurrence
  * Recurrence must be documented based on a combination of clinical and imaging parameters, consistent with routine clinical practice, with or without histologic confirmation
  * Patients may have had any number of relapses and be eligible for the study
  * Patients must have been previously treated with radiation therapy and temozolomide (bevacizumab-naïve - Groups 1 and 3) or radiation therapy, temozolomide and bevacizumab (bevacizumab-exposed -Groups 2 and 4); therapy with these agents may be given together or sequentially in the past
  * All patients may have had prior surgery, chemotherapy, and radiation therapy; prior biologic therapy is permitted only for bevacizumab-exposed patients (Groups 2 and 4); prior treatment with Gliadel is permitted for all groups
  * For bevacizumab-naïve patients (Groups 1 and 3) a minimum of 6 months must have elapsed since completion of radiation therapy for study entry, and there is no minimum time since completion of last chemotherapy; for bevacizumab-exposed patients (Groups 2 and 4) no minimum time since completion of last radiation therapy, biologic agents, or chemotherapy will be required for study entry
  * Patients must have an ECOG performance status of =< 2
  * Hemoglobin >= 10
  * Platelets >= 100,000/mm^3
  * Absolute neutrophil count >= 1500/mm^3
  * Bilirubin =< 1.5 x upper limit of normal range (ULN)
  * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 3 x ULN
  * Blood urea nitrogen (BUN) =< 1.5 x ULN
  * Creatinine =< 1.5 x ULN
  * Urine protein/creatinine ratio should be =< 1
  * Patients' baseline blood pressure must be adequately controlled with or without antihypertensive medications prior to enrollment (systolic < 140 mmHg, diastolic < 90 mmHg)
  * Patients must have a baseline evaluation including history and physical examination with neurological evaluation and magnetic resonance imaging (MRI) of the brain (with and without gadolinium-based contrast), all completed within 30 days prior to initiation of treatment
  * Female patients of child-bearing potential must have a negative pregnancy test within 14 days prior to enrollment on study; child-bearing potential is defined as any female (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets one of the following criteria:

    * Has not undergone a hysterectomy or bilateral oophorectomy
    * Or has not been naturally postmenopausal for at least 12 consecutive months (i.e. has had menses at any time in the preceding consecutive 12 months)
  * Females of child-bearing potential and sexually-active males must consent to follow acceptable birth control methods to avoid contraception while on treatment
  * All subjects must have given signed, informed consent prior to registration on study
  * Patients previously treated outside of Northwestern must have their pathology slides sent to Northwestern for review and confirmation - NOTE: a copy of the pathology report is sufficient for registration

Exclusion Criteria:

* • Patients who are pregnant or breast-feeding will NOT be eligible for participation

  • Patients with a prior malignancy will NOT be eligible for participation aside from the following exception:
* Patients who have had any curatively treated malignancy and have been disease free without treatment for 1 year prior to study entry ARE eligible for participation

  * Patients with an active second malignancy (other than non-melanoma skin cancer or cervical cancer in situ) are NOT eligible for participation
  * Patients with uncontrolled hypertension (>= 140/90 mmHg) are NOT eligible for participation
  * Patients who exhibit any other serious concurrent infection or other medical illness which would jeopardize their ability to receive the therapy outlined in this protocol with reasonable safety will NOT be eligible for participation
  * The eligibility criteria listed above are interpreted literally and cannot be waived

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2011-12-14 (Actual); Primary Completion 2018-09-12 (Actual); Study Completion 2018-09-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Raizer, MD, Principal Investigator — Northwestern University
Locations (5):
- United States (5):
  - Northwestern University, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Northwestern Lake Forest Hospital, Lake Forest, Illinois
  - Edward Cancer Center, Naperville, Illinois
  - Central Dupage Hospital, Warrenville, Illinois

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study opened for accrual on November 14, 2011 with an accrual goal of up to 77 patients and the first patient being enrolled on December 14, 2011. The study was closed permanently on March 24, 2017 due to low accrual with 54 patients treated on the study.
Groups:
- Treatment (Radiation, Chemotherapy, Monoclonal Antibody): CONCURRENT THERAPY: Patients undergo hypofractionated radiation therapy 5 days a week beginning on Day 0. Patients also receive temozolomide PO QD and bevacizumab IV over 30-90 minutes once every 2 weeks beginning on Days -3 to 0. Treatment continues for 5 weeks in the absence of disease progression or unacceptable toxicity.
  ADJUVANT THERAPY: Beginning 2 weeks after completion of radiation therapy, patients receive temozolomide PO QD for 6 weeks and bevacizumab IV over 30-90 minutes once every 2 weeks. Courses repeat every 8 weeks in the absence of disease progression or unacceptable toxicity.
  Temozolomide: Given PO
  Hypofractionated Radiation Therapy: Undergo hypofractionated radiation therapy
  Bevacizumab: Given IV
  Questionnaire administration: Ancillary studies
Period: Concurrent Therapy (5 Weeks)
Arm/Group | Treatment (Radiation, Chemotherapy, Monoclonal Antibody)
Started | 54
Completed | 38
Not Completed | 16
Not completed — Adverse Event | 4
Not completed — Death | 2
Not completed — Withdrawal by Subject | 5
Not completed — Progressive Disease | 5
Period: Started Adjuvant Therapy
Arm/Group | Treatment (Radiation, Chemotherapy, Monoclonal Antibody)
Started | 38
Completed First Cycle | 37
Completed | 37
Not Completed | 1
Not completed — Withdrawal by Subject | 1
Period: Adjuvant Therapy Until PD or Toxicity
Arm/Group | Treatment (Radiation, Chemotherapy, Monoclonal Antibody)
Started | 37
Went on to Cycle 2 + | 27
Completed | 27
Not Completed | 10
Not completed — Death | 1
Not completed — Withdrawal by Subject | 1
Not completed — Progressive Disease | 8
Period: Follow-up Until Death or 12.31.18 Occurs
Arm/Group | Treatment (Radiation, Chemotherapy, Monoclonal Antibody)
Started (All patients that receive one dose of study treatment go into the follow up portion of the study.) | 54
Completed | 54
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Radiation, Chemotherapy, Monoclonal Antibody)
Number analyzed (Participants) | 54
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 46
  >=65 years | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 37
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 48
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 3
  White | 48
  More than one race | 2
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 54
Bevacizumab-Naive Recurrent GBM [Count of Participants; unit: Participants] | 8
Bevacizumab-Exposed Recurrent GBM [Count of Participants; unit: Participants] | 36
Bevacizumab-Naive Recurrent Anaplastic Glioma [Count of Participants; unit: Participants] | 3
Bevacizumab-Exposed Recurrent Anaplastic Glioma [Count of Participants; unit: Participants] | 7

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS) for Patients With Recurrent High Grade Malignant Gliomas Treated With Concurrent Radiation, Temozolomide, and Bevacizumab Followed by Adjuvant Temozolomide and Bevacizumab.
Description: Data will be analyzed using Kaplan-Meier curves. OS is defined as the time from first re-irradiation treatment until death from any cause.
Time Frame: From treatment initiation and every 8 weeks for up to 53.5 months
Population: All patients were eligible for this outcome measure with 2 patients not experiencing the event at time of analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment (Radiation, Chemotherapy, Monoclonal Antibody)
Number analyzed (Participants) | 54
Months | 8.5 [6.4 to 9.5]

2. Secondary Outcome: Patient Reported Quality of Life (QOL)
Description: Questionnaires were completed before treatment (baseline) at the end of treatment (EOT) and after Cycle 1 and Cycle 2 of treatment (Initial phase of treatment =5 weeks + approximately 2 weeks recovery then adjuvant therapy where 1 cycle = 8 weeks). The following questionnaires were completed by patients to evaluate quality of life (QOL) at these timepoints:
  FACT-Fatigue - scores from 1 to 4 with 1=not at all and 4=very much, the higher the score the more fatigue reported by the patient.
  FACT-Brain (FACT Br) which included - Physcial Well-being (PWB), Social/Family Well-being (SWB), Emotional Well-being (EWB), and Functional Well-being (FWB).
  Patients gave scores from 0 to 4 with 0=not at all and 4=very much, the higher the score the better the QOL reported by the patient.
Time Frame: Completed before treatment (baseline) after Cycle 1 (approximately week 15) and Cycle 2 (approximately week 23)of adjuvant treatment and at the end of treatment (up to 7 cycles of adjuvant treatment, where 1 cycle =8 weeks)
Population: Only patients where sufficient data was collected for analysis were considered evaluable for this endpoint and included.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment (Radiation, Chemotherapy, Monoclonal Antibody)
Number analyzed (Participants) | 42
score on a scale
  FACT-BR Total : Baseline | 130.4 (29.6)
  FACT-BR Total : EOT | 106.9 (61.4)
  FACT-BR Total : Post Cycle 1 | 133.0 (18.8)
  FACT-BR Total : Post Cycle 2 | 131.4 (10.2)
  FACT-BR PWB : Baseline | 22.0 (5.0)
  FACT-BR PWB : EOT | 21.6 (5.0)
  FACT-BR PWB : Post Cycle 1 | 21.7 (4.4)
  FACT-BR PWB : Post Cycle 2 | 21.1 (3.9)
  FACT-BR SWB : Baseline | 22.2 (5.4)
  FACT-BR SWB : EOT | 22.9 (4.3)
  FACT-BR SWB : Post Cycle 1 | 23.0 (3.2)
  FACT-BR SWB : Post Cycle 2 | 23.7 (3.0)
  FACT-BR EWB : Baseline | 15.9 (5.7)
  FACT-BR EWB : EOT | 16.5 (4.9)
  FACT-BR EWB : Post Cycle 1 | 17.2 (3.3)
  FACT-BR EWB : Post Cycle 2 | 17.7 (3.0)
  FACT-FWB : Baseline | 15.9 (6.9)
  FACT-FWB : EOT | 17.8 (4.8)
  FACT-FWB : Post Cycle 1 | 17.0 (4.8)
  FACT-FWB: Post Cycle 2 | 18.3 (3.3)
  FACIT-Fatigue: Baseline | 35.6 (10.3)
  FACIT-Fatigue: EOT | 30.3 (12.5)
  FACIT-Fatigue: Post Cycle 1 | 34.4 (7.7)
  FACIT-Fatigue: Post Cycle 2 | 36.2 (7.9)

3. Secondary Outcome: Safety Profile for Patients With Recurrent High Grade Malignant Gliomas Treated With Concurrent Radiation, Temozolomide, and Bevacizumab Followed by Adjuvant Temozolomide and Bevacizumab
Description: Toxicity will be assessed using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 4.0 criteria on Day 1 of every treatment cycle and by patient report while on study treatment and up to 30 days after the last treatment. Grade 1 - 4 adverse events (AE) where the relationship between the AE and at least one of the study drugs were considered to be definite, probable or possible, were collected and graded as:
  Grade 1 Mild AE Grade 2 Moderate AE Grade 3 Severe AE Grade 4 Life-threatening or disabling AE Grade 5 Death related to AE
Time Frame: Completed weekly during initial phase of 5 weeks and 2 weeks recovery, then every cycle during adjuvant therapy where 1 cycle =8 weeks (for up to 7 cycles)
Population: All patients that received at least one dose of treatment on study were eligible for this outcome measure
Measure: Number; unit: participants
Arm/Group | Treatment (Radiation, Chemotherapy, Monoclonal Antibody)
Number analyzed (Participants) | 54
participants
  Lymphopenia : Grade 1 | 4
  Lymphopenia : Grade 2 | 12
  Lymphopenia : Grade 3 | 4
  Lymphopenia : Grade 4 | 1
  Fatigue : Grade 1 | 9
  Fatigue : Grade 2 | 5
  Fatigue : Grade 3 | 1
  Fatigue : Grade 4 | 0
  Thrombocytopenia : Grade 1 | 8
  Thrombocytopenia : Grade 2 | 1
  Thrombocytopenia : Grade 3 | 2
  Thrombocytopenia : Grade 4 | 1
  Anemia : Grade 1 | 7
  Anemia : Grade 2 | 1
  Anemia : Grade 3 | 1
  Anemia : Grade 4 | 0
  Constipation : Grade 1 | 8
  Constipation : Grade 2 | 1
  Constipation : Grade 3 | 0
  Constipation : Grade 4 | 0
  Hypertension : Grade 1 | 0
  Hypertension : Grade 2 | 6
  Hypertension : Grade 3 | 1
  Hypertension : Grade 4 | 0
  Neutropenia : Grade 1 | 2
  Neutropenia : Grade 2 | 3
  Neutropenia : Grade 3 | 0
  Neutropenia : Grade 4 | 0
  Epistaxis : Grade 1 | 3
  Epistaxis : Grade 2 | 0
  Epistaxis : Grade 3 | 0
  Epistaxis : Grade 4 | 0
  Thromboembolism : Grade 1 | 0
  Thromboembolism : Grade 2 | 1
  Thromboembolism : Grade 3 | 1
  Thromboembolism : Grade 4 | 0
  Proteinuria : Grade 1 | 0
  Proteinuria : Grade 2 | 0
  Proteinuria : Grade 3 | 2
  Proteinuria : Grade 4 | 0
  Wound Complication : Grade 1 | 0
  Wound Complication : Grade 2 | 0
  Wound Complication : Grade 3 | 2
  Wound Complication : Grade 4 | 0

4. Secondary Outcome: Percentage of Patients With Progression Free Survival (PFS) at 6 Months and 12 Months
Description: Progression Free Survival is defined as the time from the first study treatment to the first occurrence of disease progression or death. Data will be analyzed using Kaplan-Meier curves. Tumor measurements and assessments will be based on Updated Response Assessment Criteria of High Grade Gliomas- Neuro-Oncology Working Group (RANO criteria). Tumor assessments may include either a CT or MRI scan of the brain, however the same method should be used throughout the treatment period for each patient. In general, progressive disease is defined as any of the following: ≥ 25% increase in T1 gadolinium enhancing disease, increase in T2/Flair, new lesions present or decrease in clinical status
Time Frame: At 6 and 12 months after the start of treatment
Population: Only evaluable patients that completed RT treatment, with follow up imaging and data for progression were included in this endpoint.
Measure: Number; unit: percentage of patients with PFS
Arm/Group | Treatment (Radiation, Chemotherapy, Monoclonal Antibody)
Number analyzed (Participants) | 42
percentage of patients with PFS
  6 Months | 48
  12 Months | 12

5. Post Hoc Outcome: Response of Patients With Recurrent High Grade Malignant Gliomas Treated With Concurrent Radiation, Temozolomide, and Bevacizumab Followed by Adjuvant Temozolomide and Bevacizumab
Description: Best response is measured by CT/MRI and assessed by Updated Response Assessment Criteria of High Grade Gliomas- Neuro-Oncology Working Group (RANO criteria).
  In general best response will be defined as one of the following:
  Complete Response: No T1 gadolinium enhancing disease, stable or decreasing T2/FLAIR, no new lesions, no corticosteroid use and stable or increasing clinical status Partial Response: ≥ 50% decrease in T1 gadolinium enhancing disease, stable or decreasing T2/FLAIR, no new lesions,stable or decreasing use of corticosteroids, and stable or increasing clinical status Stable Disease: < 50% decrease but < 25% increase T1 gadolinium enhancing disease, stable or decreasing T2/FLAIR, no new lesions,stable or decreasing use of corticosteroids, and stable or increasing clinical status Progressive Disease is any of the following: ≥ 25% increase in T1 gadolinium enhancing disease, increase in T2/Flair, new lesions present or decrease in clinical status
Time Frame: Every 8 weeks from the start of study treatment. Median time from beginning of initial radiation treatment was 25.3 months (range 8.1-82.4 months)
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Radiation, Chemotherapy, Monoclonal Antibody)
Number analyzed (Participants) | 54
Participants
  Complete Response | 3
  Partial Response | 10
  Stable Disease | 28
  Progressive Disease | 9
  Not Evaluable | 4

6. Post Hoc Outcome: Median Progression Free Survival (PFS) for Patients With Recurrent High Grade Malignant Gliomas Treated With Concurrent Radiation, Temozolomide, and Bevacizumab Followed by Adjuvant Temozolomide and Bevacizumab
Description: Progression Free Survival (PFS) is defined as the time from the first study treatment to the first occurrence of disease progression or death. Data will be analyzed using Kaplan-Meier curves. Tumor measurements and assessments will be based on Updated Response Assessment Criteria of High Grade Gliomas- Neuro-Oncology Working Group (RANO criteria). Tumor assessments may include either a CT or MRI scan of the brain, however the same method should be used throughout the treatment period for each patient. In general, progressive disease is defined as any of the following: ≥ 25% increase in T1 gadolinium enhancing disease, increase in T2/Flair, new lesions present or decrease in clinical status.
Time Frame: Range from treatment initiation 0.4-26.9 months
Population: as for outcome 4
Measure: Median (Full Range); unit: Months
Arm/Group | Treatment (Radiation, Chemotherapy, Monoclonal Antibody)
Number analyzed (Participants) | 42
Months | 5.5 [0.4 to 26.9]

7. Post Hoc Outcome: Overall Survival (OS) at 6 Months and 12 Months for Patients With Recurrent High Grade Malignant Gliomas Treated With Concurrent Radiation, Temozolomide, and Bevacizumab Followed by Adjuvant Temozolomide and Bevacizumab.
Description: Data will be analyzed using Kaplan-Meier curves. OS is defined as the time from first re-irradiation treatment until death from any cause. Percentages of patients alive at that 6 months and 12 months will be calculated from the Kaplan-Meier curve.
Time Frame: At 6 and 12 months from start of treatment
Measure: Number; unit: percentage of patients alive
Arm/Group | Treatment (Radiation, Chemotherapy, Monoclonal Antibody)
Number analyzed (Participants) | 54
percentage of patients alive
  6 Months | 67
  12 Months | 28

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the first day of treatment until 30 days after the last treatment on study for up to approximately 67 weeks for any patient. Concurrent therapy was 5 weeks in length followed by 2 weeks recovery and then adjuvant therapy where 1 cycle = 8 weeks and range of cycles completed 0-7.
Arm/Group | Treatment (Radiation, Chemotherapy, Monoclonal Antibody)
All-Cause Mortality (participants affected / at risk) | 52/54
Serious Adverse Events (participants affected / at risk) | 20/54
Other Adverse Events (participants affected / at risk) | 54/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Radiation, Chemotherapy, Monoclonal Antibody) (N=54)
Anorexia (Metabolism and nutrition disorders) | 1 — Patient also with constipation, decreased urine output, impaired hearing, diploplia, dysphagia, headache, hyperglycemia, and anemia. This SAE resulted in sudden death NOS
Thromboembolic Event (Vascular disorders) | 2
Generalized Muscle Weakness (Musculoskeletal and connective tissue disorders) | 1
Muscle Weakness Right-sided (Musculoskeletal and connective tissue disorders) | 1 — Patient also with localized edema during this event
Wound Infection (Infections and infestations) | 1 — Patient also with meningitis and wound dehiscence during this event
Seizure (Nervous system disorders) | 4
Dehydration (Metabolism and nutrition disorders) | 1
Upper Respiratory Infection (Infections and infestations) | 1
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 1
Fall (Injury, poisoning and procedural complications) | 1
Depressed Level of Consciousness (Nervous system disorders) | 1 — Patient with sinus bradycardia at time of the event
Death NOS (General disorders) | 5
Platelet Count Decreased (Investigations) | 1
Hepatic Infection (Infections and infestations) | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 — Patient also with shortness of breath due to the event
Wound Complication (Injury, poisoning and procedural complications) | 1
Headache (Nervous system disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1 — Patient had a seizure at the time of the event that was thought to be due to low sodium
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Radiation, Chemotherapy, Monoclonal Antibody) (N=54)
Anemia (Blood and lymphatic system disorders) | 12
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 1
Sinus bradycardia (Cardiac disorders) | 1
Sinus tachycardia (Cardiac disorders) | 2
Ear and labyrinth disorders - Other, specify (Ear and labyrinth disorders) | 1
Ear pain (Ear and labyrinth disorders) | 1
Hearing impaired (Ear and labyrinth disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Hypothyroidism (Endocrine disorders) | 2
Blurred vision (Eye disorders) | 9
Dry eye (Eye disorders) | 1
Extraocular muscle paresis (Eye disorders) | 1
Eye disorders - Other, specify (Eye disorders) | 2
Watering eyes (Eye disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Anal hemorrhage (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 21
Diarrhea (Gastrointestinal disorders) | 3
Dry mouth (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 3
Dysphagia (Gastrointestinal disorders) | 2
Esophagitis (Gastrointestinal disorders) | 1
Fecal incontinence (Gastrointestinal disorders) | 3
Gastroesophageal reflux disease (Gastrointestinal disorders) | 4
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1
Mucositis oral (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 14
Oral pain (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 6
Chills (General disorders) | 1
Edema limbs (General disorders) | 2
Fatigue (General disorders) | 31
Fever (General disorders) | 1
Gait disturbance (General disorders) | 15
Infusion site extravasation (General disorders) | 1
Irritability (General disorders) | 2
Localized edema (General disorders) | 2
Malaise (General disorders) | 1
Pain (General disorders) | 6
Sudden death NOS (General disorders) | 1
Immune system disorders - Other, specify (Immune system disorders) | 1
Infections and infestations - Other, specify (Infections and infestations) | 2
Meningitis (Infections and infestations) | 1
Peripheral nerve infection (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Tooth infection (Infections and infestations) | 1
Upper respiratory infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 2
Bruising (Injury, poisoning and procedural complications) | 1
Dermatitis radiation (Injury, poisoning and procedural complications) | 7
Fall (Injury, poisoning and procedural complications) | 3
Fracture (Injury, poisoning and procedural complications) | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 4
Alkaline phosphatase increased (Investigations) | 2
Aspartate aminotransferase increased (Investigations) | 6
Blood bilirubin increased (Investigations) | 3
Cholesterol high (Investigations) | 2
Creatinine increased (Investigations) | 3
INR increased (Investigations) | 1
Investigations - Other, specify (Investigations) | 1
Lymphocyte count decreased (Investigations) | 27
Lymphocyte count increased (Investigations) | 1
Neutrophil count decreased (Investigations) | 2
Platelet count decreased (Investigations) | 20
Urine output decreased (Investigations) | 1
Weight gain (Investigations) | 3
Weight loss (Investigations) | 10
White blood cell decreased (Investigations) | 10
Anorexia (Metabolism and nutrition disorders) | 11
Dehydration (Metabolism and nutrition disorders) | 5
Hyperglycemia (Metabolism and nutrition disorders) | 14
Hyperkalemia (Metabolism and nutrition disorders) | 1
Hypertriglyceridemia (Metabolism and nutrition disorders) | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 8
Hypocalcemia (Metabolism and nutrition disorders) | 8
Hypoglycemia (Metabolism and nutrition disorders) | 3
Hypokalemia (Metabolism and nutrition disorders) | 5
Hypomagnesemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 3
Back pain (Musculoskeletal and connective tissue disorders) | 1
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1
Joint range of motion decreased cervical spine (Musculoskeletal and connective tissue disorders) | 1
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 7
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 3
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 7
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4
Akathisia (Nervous system disorders) | 1
Amnesia (Nervous system disorders) | 2
Ataxia (Nervous system disorders) | 8
Cognitive disturbance (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 5
Dysarthria (Nervous system disorders) | 3
Dysgeusia (Nervous system disorders) | 2
Dysphasia (Nervous system disorders) | 13
Edema cerebral (Nervous system disorders) | 7
Encephalopathy (Nervous system disorders) | 1
Facial nerve disorder (Nervous system disorders) | 6
Headache (Nervous system disorders) | 20
Hypersomnia (Nervous system disorders) | 1
Lethargy (Nervous system disorders) | 2
Memory impairment (Nervous system disorders) | 11
Movements involuntary (Nervous system disorders) | 1
Nervous system disorders - Other, specify (Nervous system disorders) | 9
Paresthesia (Nervous system disorders) | 5
Peripheral sensory neuropathy (Nervous system disorders) | 4
Presyncope (Nervous system disorders) | 1
Pyramidal tract syndrome (Nervous system disorders) | 7
Seizure (Nervous system disorders) | 20
Somnolence (Nervous system disorders) | 2
Stroke (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 5
Anxiety (Psychiatric disorders) | 13
Confusion (Psychiatric disorders) | 9
Depression (Psychiatric disorders) | 13
Hallucinations (Psychiatric disorders) | 2
Insomnia (Psychiatric disorders) | 10
Personality change (Psychiatric disorders) | 2
Psychiatric disorders - Other, specify (Psychiatric disorders) | 1
Psychosis (Psychiatric disorders) | 1
Chronic kidney disease (Renal and urinary disorders) | 1
Hematuria (Renal and urinary disorders) | 1
Proteinuria (Renal and urinary disorders) | 6
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 2
Urinary frequency (Renal and urinary disorders) | 1
Urinary incontinence (Renal and urinary disorders) | 7
Urinary retention (Renal and urinary disorders) | 2
Urinary tract pain (Renal and urinary disorders) | 1
Urinary urgency (Renal and urinary disorders) | 3
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 4
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 3
Alopecia (Skin and subcutaneous tissue disorders) | 16
Nail loss (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2
Purpura (Skin and subcutaneous tissue disorders) | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 20
Thromboembolic event (Vascular disorders) | 4

LIMITATIONS AND CAVEATS:
The study was closed to accrual before the accrual goal was met due to slow accrual

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-28): https://cdn.clinicaltrials.gov/large-docs/21/NCT01478321/Prot_SAP_000.pdf